CLINICAL TRIAL: NCT03892512
Title: The Effect of Dexmedetomidine and Esmolol on Early Post Operative Cognitive Dysfunction After Middle Ear Surgery Under Hypotensive Technique :Comparative , Randomized Double Blinded Study
Brief Title: Dexmedetomidine and Esmolol Early Post Operative Cognitive Dysfunction
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Samaa Rashwan, Samaa Abou Alkassem Rashwan, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Beni-Suef
Record Dates: First submitted 2019-03-23; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — esmolol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomedine (Active Comparator): The Patients will receive hypotensive anesthesia via I .V infusion with dexmedetomidine (Percedex .Pfizer CO ) .
  Interventions: Drug: Dexmedetomidine
- esmolol (Active Comparator): Patients will receive hypotensive anesthesia via I .V infusion with esmolol ( Esmolol Hydrochloride . Baxter CO ).
  Interventions: Drug: Esmolol Hydrochloride

INTERVENTIONS:
Drug: Esmolol Hydrochloride — Patients will receive hypotensive anesthesia via I .V infusion with esmolol ( Esmolol Hydrochloride )
  Other Names: esmolol
  Arms: esmolol
Drug: Dexmedetomidine — The Patients will receive hypotensive anesthesia via I .V infusion with dexmedetomidine (Percedex )
  Other Names: precedex
  Arms: dexmedetomedine

SUMMARY:
Dexmedetomidine is a highly selective α2adrenoceptor agonist recently introduced to anesthesia that produces dose dependent sedation, anxiolysis, and analgesia (involving spinal and supraspinal sites) without respiratory depression.

From a pharmacokinetic perspective,dexmedetomidine has a half life of nearly 2 hours, duration of action of nearly 4 hour, and thus, a side effect profile that is shorter in duration than clonidine.

Esmolol is a cardioselective beta₁ receptor blocker with rapid onset, a very short duration of action (elimination half-life is approximately 9 minutes) , and no significant intrinsic sympathomimetic or membrane stabilising activity at therapeutic dosages

DETAILED DESCRIPTION:
The study will be a randomized double blinded study and will be carried by the Department of Anaesthesia at Beni-Suef University Hospital after obtaining approval from local research and ethical committee. Written informed consent will be obtained from each patient before operation. Aiming to assess of the early cognitive dysfunction after controlled hypotensive anesthesia with either dexmedetomidine or esmolol during middle ear surgeries

ELIGIBILITY:
Inclusion Criteria:

Patients aging 20-50 years ASA physical status I-II . Males , females

Exclusion Criteria:

1. hypertensive patient
2. Patients receiving sedatives as midazolam.
3. Patients with ischemic heart diseases, heart block, congestive heart failure, valvular heart diseases.
4. Patients with cerebrovascular diseases.
5. Patients with impaired kidney function.
6. Patients with history of chronic liver diseases.
7. Patients with asthma, chronic obstructive lung diseases.
8. Patients with diabetes mellitus, coagulation disorders, pregnancy.
9. Patients with history of allergy to the drugs used in the study or patients with substance abuse .

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
assess the early cognitive dysfunction after controlled hypotensive anesthesia | MMS will performed at 1 hour, 6 and 24 hours postoperatively .The mximum score will be 30 points, a decrease of 2 or more will be considered as cognitive function decline. score less than 23 will be considered as cognitive impairmen
  mini mental state examination (MMSE) will be used for evaluation of cognitive function Data will be expressed in mean ± SD and were compared using analysis of variance (ANOVA). The significance of non-parametric data was determined using chi-square test. For all comparisons P < 0.05 was considered significant.,

CONTACTS AND LOCATIONS:
Overall Officials: Samaa ak Rashwan, MD, Principal Investigator — Assisstant proffesor of anesthesia
Locations (1):
- Beni-Suef University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided